CLINICAL TRIAL: NCT02417675
Title: Postpartum Adherence Clubs to Enhance Support: the PACER Study
Acronym: PACER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Elaine J. Abrams, MD, Senior Research Director, ICAP, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AAAO5601; 3R01HD074558-03S1 (NIH)
Record Dates: First submitted 2015-04-01; First posted 2015-04-16 (Estimated); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: HIV
Keywords: Option B+; Adherence Club; Postpartum; Breastfeeding; Mother-to-child transmission
MeSH Terms: conditions — Breast Feeding | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard of Care (SOC) (Active Comparator): Women who choose the SOC will receive postpartum antiretroviral therapy (ART) services at their nearest primary care clinic, following the Standard of Care for Mothers. Details are provided in the intervention description.
  Infants receive the same care in each arm, according to the Standard of Care for Infants.
  Interventions: Other: Standard of Care for Mothers; Other: Standard of Care for Infants
- Intervention (AC) (Experimental): Women who choose the Community-based Adherence Clubs (AC) will receive postpartum antiretroviral therapy (ART) services at an AC, rather than at their nearest primary care clinic as in the SOC arm. Details are provided in the intervention section.
  Infants receive the same care in each arm, according to the Standard of Care for Infants.
  Interventions: Other: Community-based Adherence Clubs; Other: Standard of Care for Infants

INTERVENTIONS:
Other: Community-based Adherence Clubs — Women in the AC arm are prescribed 2 months of their current ART medication (compared to 1 month in the SOC) and will be advised to go to the AC office immediately, where they will be scheduled for their first session. Women will attend AC meetings every two months. At these meetings, women will receive a 2 month supply of medication, health education and peer-support. A trained Community Health Worker (CHW) will also collect blood samples, weight, and current signs/symptoms from women.
  Each participant has 5 working days after their AC session to come and collect her medication. Those who have defaulted will be followed up by the CHW via phone calls and, possibly, home visits. If reached, women will be told to return immediately to the main ART facility for receipt of ART care.
  Other Names: AC
  Arms: Intervention (AC)
Other: Standard of Care for Mothers — Women will be referred immediately from the maternity ART clinic to their nearest adult ART clinic at their first postpartum clinic visit. At referral, they receive an initial 1-month supply of their current ART medication. At the first appointment after transfer into the general ART service, patients undergo clinical history and examination by a doctor or clinical nurse practitioner. Laboratory investigations are ordered according to standard protocols or based on clinician discretion. For the 1st 4 months in the new service, stable patients are dispensed 1 month of ART; subsequent visits are 2-monthly for medication refill, with clinician review 6-monthly; patients with particular clinical or psychosocial concerns may be reviewed more regularly, or referred to higher levels of care.
  Other Names: SOC
  Arms: Standard of Care (SOC)
Other: Standard of Care for Infants — All infants will receive care at their nearest primary care clinic. Following national protocols, all HIV-infected mothers are issued a 6-week supply of nevirapine syrup after delivery and counselled on daily nevirapine prophylaxis. Infant follow-up takes place within 1 week postpartum with the mother (at the MOU) and then at 6 weeks postpartum (at the nearest primary care clinic) when HIV PCR testing of the infant is carried out. Following national protocols, infants who are breastfed beyond 6 weeks receive HIV PCR testing 2-4 weeks after the cessation of breastfeeding, again conducted at the nearest City of Cape Town primary care clinic.

SUMMARY:
The Western Cape province of South Africa (SA) is changing the way it treats pregnant women with HIV. Now, all HIV-infected pregnant women, regardless of how sick or healthy they are, will receive antiretroviral treatment (ART) for life ("Option B+"). However, there are few well-developed models of service delivery to support this change to "Option B+" in the Western Cape and many parts of the continent.

The parent study -- Strategies to Optimize ART Services for Maternal & Child Health (MCH-ART)-- is testing two clinic-based models of service delivery for Option B+ . To complement MCH-ART, this study, PACER, will test whether community-based Adherence Clubs are an effective model for keeping breastfeeding women in HIV care after pregnancy. These clubs have been used to free up space at ART clinics by moving stable HIV+ patients to community-based services, but they have not been studied as an effective strategy among breastfeeding women after delivery. PACER seeks to address this gap.

DETAILED DESCRIPTION:
The Western Cape province of South Africa (SA) is implementing the policy of universal initiation of lifelong ART in all HIV-infected pregnant women regardless of CD4 cell count or disease stage ("Option B+"). However there are few well-developed models of service delivery to support implementation of "Option B+" in the Western Cape and many parts of the continent. In particular, while systems for initiation and follow-up of pregnant women on ART are based within well-established antenatal care clinics (ANC), there are major concerns regarding delivery of ART to HIV-infected women during the postpartum period. Multiple studies indicate high levels of non-retention in care, and/or inadequate ART adherence, during the postpartum period, presenting a threat to HIV-infected women and their infants.4-8 In turn, there is an urgent need for evidence-based approaches to support the growing number of HIV-infected mothers on ART.

In this context, the parent study-- Strategies to Optimize ART Services for Maternal & Child Health (MCH-ART)-- provides a rigorous implementation science framework for understanding optimal approaches for managing HIV-infected women and their HIV-exposed infants in the first year after delivery under "Option B+". While MCH-ART focuses on clinic-based models of care, there is also growing attention to the role of community health workers (CHWs) in supporting patients on ART, including community-based distribution and adherence support away from health facilities.To complement MCH-ART, the PACER study aims to investigate community-based Adherence Clubs as an effective model for engaging and retaining breastfeeding women beyond pregnancy to maximize maternal and infant health. In Cape Town, specifically, Adherence Clubs have been developed in which ART services are located away from clinics and are led by CHWs with support from ART clinic nurses. These clubs have been implemented to help decongest ART clinics by shifting stable patients to community-based services, but they have not been studied as an effective strategy among breastfeeding women in the postpartum period. PACER seeks to address this gap by randomizing women in the parent study, MCH-ART, to either the AC system or to the nearest adult ART clinic. Infants in both arms will receive the same services, following the local standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Documented HIV-infection according to two finger-prick rapid tests using different test types (per routine protocol in this setting) or documentation of HIV status for those women self reporting HIV diagnosis.
* Initiated ART during the antenatal period (during most recent pregnancy)
* Within one month postpartum
* Currently breastfeeding within one month postpartum
* Willingness to return for postnatal study visits
* Able to provide informed consent for research
* Eligible to receive care at local Adherence Club, based on following local eligibility criteria:

  1. Virally suppressed (HIV RNA <1000 copies/mL) per most recent viral load test (conducted during pregnancy)
  2. Clinically stable (no active co-morbidity including opportunistic infections)
  3. Current resident of a catchment area appropriate for Adherence Club referral
* Infants of women enrolled in the study.

Exclusion Criteria:

* Receipt of any ART services outside the Gugulethu MOU ART service in the postpartum period
* Intention to relocate out of Cape Town permanently during the following one year
* Any medical, psychiatric or social condition which in the opinion of the investigators would affect the ability to consent and/or participate in the study, including:

  1. Refusal to take ART/ARVs
  2. Denial of HIV status

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2015-02; Primary Completion 2016-10-31 (Actual); Study Completion 2016-10-31 (Actual)

PRIMARY OUTCOMES:
Maternal retention | 12 months
  Proportion of mothers retained in HIV care and adhering to ART at 12 months postpartum

SECONDARY OUTCOMES:
Maternal Loss to Follow-up | 12 months
  Proportion of women who are lost to follow-up on ART at 12 months postpartum.
Maternal Viral Suppression | 12 months
  Proportion of women with viral suppression at the end of the breastfeeding period.
Infant HIV diagnosis | 12 months
  Proportion of infants receiving proper HIV diagnosis at 12 months postpartum
Infant vaccination | 12 months
  Proportion of infants receiving proper vaccinations at 12 months postpartum
Mother-to-child transmission | 12 months
  Rate of HIV transmission from mother-to-child

CONTACTS AND LOCATIONS:
Overall Officials: Elaine J Abrams, MD, Principal Investigator — ICAP at Columbia University; Landon Myer, MD, Principal Investigator — University of Cape Town
Locations (1):
- Gugulethu Community Health Centre, Cape Town, Western Cape, South Africa

REFERENCES:
- [Derived] Zerbe A, Brittain K, Phillips TK, Iyun VO, Allerton J, Nofemela A, Kalombo CD, Myer L, Abrams EJ. Community-based adherence clubs for postpartum women on antiretroviral therapy (ART) in Cape Town, South Africa: a pilot study. BMC Health Serv Res. 2020 Jul 8;20(1):621. doi: 10.1186/s12913-020-05470-5. PMID 32641032
- [Derived] Trafford Z, Gomba Y, Colvin CJ, Iyun VO, Phillips TK, Brittain K, Myer L, Abrams EJ, Zerbe A. Experiences of HIV-positive postpartum women and health workers involved with community-based antiretroviral therapy adherence clubs in Cape Town, South Africa. BMC Public Health. 2018 Jul 31;18(1):935. doi: 10.1186/s12889-018-5836-4. PMID 30064405